CLINICAL TRIAL: NCT05908513
Title: Randomized Study on N-acetylcysteine Treatment and Outcomes in Patients With Advanced Atherosclerotic Heart Diseases and Diabetes Mellitus (RENEWAL)
Brief Title: NAC Treatment and Outcomes in Patients With Advanced Atherosclerosis and DM
Acronym: RENEWAL
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Lack of available resources needed to conduct study.
Sponsor: University of Missouri-Columbia (Other)
Collaborators: Shandong Provincial Hospital (Other Government); Central South University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2072662
Record Dates: First submitted 2021-10-04; First posted 2023-06-18 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Atherosclerosis of Artery; Peripheral Artery Disease; Diabetes Mellitus; Inflammation; Oxidative Stress
Keywords: Atherosclerosis, ROS, Inflammation, Diabetes
MeSH Terms: conditions — Peripheral Arterial Disease; Diabetes Mellitus; Inflammation; Atherosclerosis | interventions — Acetylcysteine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: We will use double blind for this study. Neither the participants nor the researcher knows which treatment or intervention participants are receiving until the clinical trial is over.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- NAC treatment (Active Comparator): N-acetylcysteine capsule, 600mg/day, oral, 5 years
  Interventions: Drug: N-acetylcysteine
- Placebo (Placebo Comparator): Similar chemical structure of NAC but without function
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: N-acetylcysteine — Will be used as capsule form, 600mg per day if the patient can tolerate it. If not, we may decrease the dosage.
  Other Names: Acetadote
  Arms: NAC treatment
Drug: Placebo — Similar chemical structure of NAC but without function
  Arms: Placebo

SUMMARY:
Atherosclerosis and diabetes are related to coronary artery disease and peripheral artery disease. The mechanisms are related to increased reactive oxygen species (ROS) formation and inflammatory cytokine secretion. However, simply using antioxidant or anti-inflammatory therapies has no optimal outcomes. On the other hand, N-acetylcysteine (NAC) which has both antioxidant and anti-inflammatory effects could effectively attenuate ROS production and reduce vascular inflammation. Hence, we will investigate the effect of NAC treatment on the outcomes in patients with advanced atherosclerotic heart diseases and patients with diabetes combined with significant peripheral artery disease.

DETAILED DESCRIPTION:
Atherosclerosis is a chronic inflammatory disease and remains one of the major causes of death globally, despite aggressive risk stratifications including smoking cessation, optimal control of lipid, blood pressure, and diabetes. Antioxidant therapies with vitamin E and C or β-carotene failed to achieve significant clinical benefits in patients with cardiovascular diseases (CVD) including atherosclerosis. New therapies including interleukin-1β monoclonal antibody canakinumab and anti-inflammatory drug colchicine could significantly reduce the rate of major adverse cardiovascular events (MACE) including nonfatal myocardial infarction, nonfatal stroke, or cardiovascular death. However, canakinumab therapy did not decrease all-cause mortality, and was associated with a significant increase in the incidence of fatal infection (including sepsis), and high cost. While colchicine is a generic drug and decreases the rate of MACE, colchicine therapy is associated with a significant increase in death from non-cardiovascular causes5. Thus, alternative options are needed to attenuate atherosclerosis. N-acetylcysteine (NAC) has been traditionally considered an antioxidant although it is more like an anti-inflammatory agent, and could effectively attenuate reactive oxygen species (ROS) production, and reduce vascular inflammation. NAC significantly decreases the progression of atherosclerosis in young apolipoprotein E-deficient mice and low-density lipoprotein receptor deficient (LDLR-/-) mice with an atherogenic high fat diet (HFD). NAC treatment delays cellular senescence in endothelial cells from atherosclerotic patients, and improves coronary and peripheral endothelium-dependent vasodilation in human subjects with or without atherosclerosis. NAC treatment also inhibits oxidized LDL-induced foam cell formation and suppresses matrix-degrading capacity of foam cells. However, it is unclear if NAC could attenuate the progression of atherosclerosis or reverse the course of atherosclerosis in aging mice. Diabetes mellitus (DM) significantly increases the risk of developing severe peripheral artery disease (PAD) with critical limb ischemia (CLI) and chronic ulcers. Due to poor healing, patients with diabetic CLI may need limb amputation that accounts for about 60% of all non-traumatic amputations in the U. S. After a two decade reduction in diabetes-related non-traumatic lower-extremity amputation, recent data show an increase in amputation, particularly in young and middle-aged adults. In addition, major randomized clinical trials have shown that blood glucose-lowering or anti-hypertensive therapies have very limited effects on reducing macrovascular complications, and no benefit on amputation rates in diabetic patients. These highlight an urgent need for alterative effective approaches to promoting the recovery of diabetic ischemic limb to reduce lower-extremity amputation in DM. It is known that reactive oxygen species (ROS) production and oxidative stress are significantly increased in DM, and excessive oxidative stress is closely involved in the development of diabetic complications, including cardiovascular diseases, nephropathy, and retinopathy. Although low levels of ROS function as signaling molecules to mediate various biological responses such as gene expression, cell proliferation, migration, angiogenesis, apoptosis, and senescence in endothelial cells (ECs), high levels of ROS could contribute to a variety of pathologic conditions, including reduced nitric oxide (NO) bioavailability, impairment of vascular function and other endothelial phenotypic abnormalities. The metabolic abnormalities in DM could cause mitochondrial superoxide overproduction in endothelial cells of both large and small vessels, as well as in the myocardium. Increased glucose levels could stimulate ROS production, leading to further glucose uptake and triggering cell toxicity and death. In addition, increased formation of advanced glycation end-products (AGEs) could enhance the activity of ROS-generating enzymes including NADPH oxidase, exacerbating oxidative stress and mitochondrial superoxide production. Thus, the objectives of the proposed study are: 1) to investigate the effect of NAC treatment on the outcomes in patients with advanced atherosclerotic heart diseases and not a candidate for revascularization; and 2) to investigate the effect of NAC treatment on the outcomes in diabetic patients with significant peripheral artery disease.

ELIGIBILITY:
Inclusion Criteria:

* 1) significant coronary artery disease (CAD) and not a candidate for revascularization (CABG or PCI), or 2) significant peripheral artery disease (PAD) with or without critical limb ischemia (CLI) or chronic ulcers.

Exclusion Criteria:

* 1) Pregnant or nursing (lactating) women, confirmed by a positive hCG laboratory test 2). Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, UNLESS they are a. Women are considered post-menopausal and not of child bearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g. age appropriate, history of vasomotor symptoms) or have had surgical bilateral oophorectomy (with or without hysterectomy) or tubal ligation at least six weeks ago. In the case of oophorectomy alone or partial or total hysterectomy, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment is she considered not of child bearing potential.

  3). Planned coronary revascularization (PCI or CABG) or any other major surgical procedure.

  4). Major non-cardiac surgical or major endoscopic procedure within the past 6 months prior to the initial visit (Visit 1) 5). Multi-vessel CABG surgery within the past 3 years 6). Symptomatic patients with Class IV heart failure (HF) (New York Heart Association).

  7). Uncontrolled hypertension (defined as an average SBP >180 mmHg or an average diastolic blood pressure (DBP) >110 mmHg at Visit 1. Patients are allowed to be re-evaluated, at the discretion of investigator for this criterion if anti-hypertensive therapy has been started or increased as a result of initial screening blood pressure above these limits.

  8). Uncontrolled diabetes with persistent fasting blood glucose level of 300 or A1C of 7.5 for 3 months or defined by the investigator 9). Kidney or other organ transplant (due to anti-immune therapy) at Visit 1 10). Prior malignancy other than basal cell skin carcinoma. 11). A history of alcohol and/or substance abuse that could interfere with the conduct of the trial.

  12). History of ongoing, chronic or recurrent infectious disease except hepatitis.

  13). History of hypersensitivity to NAC. 14). Patients who have received an investigational drug or device within 30 days (inclusive) of Visit 1, or who are expected to participate in any other investigational drug or device study during the conduct of this trial, except for patients who have an investigational drug eluting stent (DES), provided that they have completed the DES trial. FDA/country-specific drug regulatory authority approved DES devices are permitted.

  15). Any life threatening condition with life expectancy < 3 years, other than vascular disease that might prevent the patient from completing the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-10-15 (Actual); Primary Completion 2021-10-15 (Actual); Study Completion 2021-10-15 (Actual)

PRIMARY OUTCOMES:
Change of blood pressure over time points | baseline, 3 months, 6 months, and 12 months
  Diastolic and systolic blood pressure
Change of biomarkers over time points | baseline, 3 months, 6 months, and 12 months
  Blood samples (5ml) will be taken for biomarkers analysis (complete blood cell count [CBC], biochemistry, Thyroid stimulating hormone [TSH], renal function, C-reactive protein [CRP], IL-1β, IL-6, TNF-α, and lipids profiles).
Change of heart rate over time points | 1 baseline, 3 months, 6 months, and 12 months
  Number of beats per minute
Change of body weight over time points | baseline, 3 months, 6 months, and 12 months
  Measured in kg

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - Shandong Provincial Hospital, Jinan, Shandong

IPD SHARING:
Plan to Share IPD: No
Due to the confidential information included in this study, all data won't be shared for now.

REFERENCES:
- [Background] Virani SS, Alonso A, Benjamin EJ, Bittencourt MS, Callaway CW, Carson AP, Chamberlain AM, Chang AR, Cheng S, Delling FN, Djousse L, Elkind MSV, Ferguson JF, Fornage M, Khan SS, Kissela BM, Knutson KL, Kwan TW, Lackland DT, Lewis TT, Lichtman JH, Longenecker CT, Loop MS, Lutsey PL, Martin SS, Matsushita K, Moran AE, Mussolino ME, Perak AM, Rosamond WD, Roth GA, Sampson UKA, Satou GM, Schroeder EB, Shah SH, Shay CM, Spartano NL, Stokes A, Tirschwell DL, VanWagner LB, Tsao CW; American Heart Association Council on Epidemiology and Prevention Statistics Committee and Stroke Statistics Subcommittee. Heart Disease and Stroke Statistics-2020 Update: A Report From the American Heart Association. Circulation. 2020 Mar 3;141(9):e139-e596. doi: 10.1161/CIR.0000000000000757. Epub 2020 Jan 29. PMID 31992061
- [Background] Bjelakovic G, Nikolova D, Gluud LL, Simonetti RG, Gluud C. Mortality in randomized trials of antioxidant supplements for primary and secondary prevention: systematic review and meta-analysis. JAMA. 2007 Feb 28;297(8):842-57. doi: 10.1001/jama.297.8.842. PMID 17327526
- [Background] Thompson PL, Nidorf SM. Colchicine: an affordable anti-inflammatory agent for atherosclerosis. Curr Opin Lipidol. 2018 Dec;29(6):467-473. doi: 10.1097/MOL.0000000000000552. PMID 30320614
- [Background] Ridker PM, Everett BM, Thuren T, MacFadyen JG, Chang WH, Ballantyne C, Fonseca F, Nicolau J, Koenig W, Anker SD, Kastelein JJP, Cornel JH, Pais P, Pella D, Genest J, Cifkova R, Lorenzatti A, Forster T, Kobalava Z, Vida-Simiti L, Flather M, Shimokawa H, Ogawa H, Dellborg M, Rossi PRF, Troquay RPT, Libby P, Glynn RJ; CANTOS Trial Group. Antiinflammatory Therapy with Canakinumab for Atherosclerotic Disease. N Engl J Med. 2017 Sep 21;377(12):1119-1131. doi: 10.1056/NEJMoa1707914. Epub 2017 Aug 27. PMID 28845751
- [Background] Nidorf SM, Fiolet ATL, Mosterd A, Eikelboom JW, Schut A, Opstal TSJ, The SHK, Xu XF, Ireland MA, Lenderink T, Latchem D, Hoogslag P, Jerzewski A, Nierop P, Whelan A, Hendriks R, Swart H, Schaap J, Kuijper AFM, van Hessen MWJ, Saklani P, Tan I, Thompson AG, Morton A, Judkins C, Bax WA, Dirksen M, Alings M, Hankey GJ, Budgeon CA, Tijssen JGP, Cornel JH, Thompson PL; LoDoCo2 Trial Investigators. Colchicine in Patients with Chronic Coronary Disease. N Engl J Med. 2020 Nov 5;383(19):1838-1847. doi: 10.1056/NEJMoa2021372. Epub 2020 Aug 31. PMID 32865380
- [Background] Salamon S, Kramar B, Marolt TP, Poljsak B, Milisav I. Medical and Dietary Uses of N-Acetylcysteine. Antioxidants (Basel). 2019 Apr 28;8(5):111. doi: 10.3390/antiox8050111. PMID 31035402
- [Background] Voghel G, Thorin-Trescases N, Farhat N, Mamarbachi AM, Villeneuve L, Fortier A, Perrault LP, Carrier M, Thorin E. Chronic treatment with N-acetyl-cystein delays cellular senescence in endothelial cells isolated from a subgroup of atherosclerotic patients. Mech Ageing Dev. 2008 May;129(5):261-70. doi: 10.1016/j.mad.2008.01.004. Epub 2008 Jan 20. PMID 18302967
- [Background] Sung HJ, Kim J, Kim Y, Jang SW, Ko J. N-acetyl cysteine suppresses the foam cell formation that is induced by oxidized low density lipoprotein via regulation of gene expression. Mol Biol Rep. 2012 Mar;39(3):3001-7. doi: 10.1007/s11033-011-1062-1. Epub 2011 Jun 17. PMID 21681422
- [Background] Anderson JL, Halperin JL, Albert NM, Bozkurt B, Brindis RG, Curtis LH, DeMets D, Guyton RA, Hochman JS, Kovacs RJ, Ohman EM, Pressler SJ, Sellke FW, Shen WK. Management of patients with peripheral artery disease (compilation of 2005 and 2011 ACCF/AHA guideline recommendations): a report of the American College of Cardiology Foundation/American Heart Association Task Force on Practice Guidelines. Circulation. 2013 Apr 2;127(13):1425-43. doi: 10.1161/CIR.0b013e31828b82aa. Epub 2013 Mar 1. No abstract available. PMID 23457117
- [Background] Hoffstad O, Mitra N, Walsh J, Margolis DJ. Diabetes, lower-extremity amputation, and death. Diabetes Care. 2015 Oct;38(10):1852-7. doi: 10.2337/dc15-0536. Epub 2015 Jul 22. PMID 26203063
- [Background] Geiss LS, Li Y, Hora I, Albright A, Rolka D, Gregg EW. Resurgence of Diabetes-Related Nontraumatic Lower-Extremity Amputation in the Young and Middle-Aged Adult U.S. Population. Diabetes Care. 2019 Jan;42(1):50-54. doi: 10.2337/dc18-1380. Epub 2018 Nov 8. PMID 30409811
- [Background] Malik RA, Tesfaye S, Ziegler D. Medical strategies to reduce amputation in patients with type 2 diabetes. Diabet Med. 2013 Aug;30(8):893-900. doi: 10.1111/dme.12169. PMID 23445087
- [Background] Howangyin KY, Silvestre JS. Diabetes mellitus and ischemic diseases: molecular mechanisms of vascular repair dysfunction. Arterioscler Thromb Vasc Biol. 2014 Jun;34(6):1126-35. doi: 10.1161/ATVBAHA.114.303090. Epub 2014 Mar 27. PMID 24675660
- [Background] Forrester SJ, Kikuchi DS, Hernandes MS, Xu Q, Griendling KK. Reactive Oxygen Species in Metabolic and Inflammatory Signaling. Circ Res. 2018 Mar 16;122(6):877-902. doi: 10.1161/CIRCRESAHA.117.311401. PMID 29700084
- [Background] Giacco F, Brownlee M. Oxidative stress and diabetic complications. Circ Res. 2010 Oct 29;107(9):1058-70. doi: 10.1161/CIRCRESAHA.110.223545. PMID 21030723
- [Background] Singh DK, Winocour P, Farrington K. Oxidative stress in early diabetic nephropathy: fueling the fire. Nat Rev Endocrinol. 2011 Mar;7(3):176-84. doi: 10.1038/nrendo.2010.212. Epub 2010 Dec 14. PMID 21151200
- [Background] Arden GB, Sivaprasad S. Hypoxia and oxidative stress in the causation of diabetic retinopathy. Curr Diabetes Rev. 2011 Sep;7(5):291-304. doi: 10.2174/157339911797415620. PMID 21916837
- [Background] Frey RS, Ushio-Fukai M, Malik AB. NADPH oxidase-dependent signaling in endothelial cells: role in physiology and pathophysiology. Antioxid Redox Signal. 2009 Apr;11(4):791-810. doi: 10.1089/ars.2008.2220. PMID 18783313
- [Background] Incalza MA, D'Oria R, Natalicchio A, Perrini S, Laviola L, Giorgino F. Oxidative stress and reactive oxygen species in endothelial dysfunction associated with cardiovascular and metabolic diseases. Vascul Pharmacol. 2018 Jan;100:1-19. doi: 10.1016/j.vph.2017.05.005. Epub 2017 Jun 1. PMID 28579545
- [Background] Liemburg-Apers DC, Willems PH, Koopman WJ, Grefte S. Interactions between mitochondrial reactive oxygen species and cellular glucose metabolism. Arch Toxicol. 2015 Aug;89(8):1209-26. doi: 10.1007/s00204-015-1520-y. Epub 2015 Jun 6. PMID 26047665
- [Background] Kunkemoeller B, Kyriakides TR. Redox Signaling in Diabetic Wound Healing Regulates Extracellular Matrix Deposition. Antioxid Redox Signal. 2017 Oct 20;27(12):823-838. doi: 10.1089/ars.2017.7263. Epub 2017 Aug 10. PMID 28699352